CLINICAL TRIAL: NCT04309838
Title: LENUS Pro® Study (LPS-II) - Observation Study With Implantable Medication Pump for Intravenous REMODULIN® (Treprostinil) Therapy in Patients With Pulmonary Arterial Hypertension
Brief Title: Observation Study With Implantable Medication Pump for Intravenous Treprostinil Therapy in Patients With Pulmonary Arterial Hypertension
Acronym: LPS-II
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: OMT GmbH & Co. KG (Unknown)
Responsible Party: Sponsor
Other Study IDs: LPS-II
Record Dates: First submitted 2020-02-20; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Arterial Hypertension; PAH
Keywords: PAH; Pulmonary arterial hypertension; Treprostinil
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Treprostinil via implanted pump — Patients, diagnosed with PAH classified in stagnating intermediate-risk status after triple therapy including Selexipag for at least three months will receive the implantation of LENUS pro that enables permanent infusion of Treprostinil.

SUMMARY:
The study is designed as a non-interventional, multicenter, prospective single-arm study to observe the therapy with REMODULIN (Treprostinil) applicated by an implantable pump in patients with pulmonary arterial hypertension (PAH).

DETAILED DESCRIPTION:
Patients that suffer from progressing PAH are medicated with intravenous prostanoids since the 80's of the last century. Nowadays, specific treatment of PAH can be realized by the huge number of substances that are currently available. Still, the time point of starting an intravenous medication is not defined yet. By evaluation of data concerning risk strata of PAH patients, this issue may be enlightened properly.

Previously collected data concerning risk-adapted therapy in PAH-patient have shown that the mortality is little in the "low-risk-status" patients, only. Thus, all efforts must be undertaken to define the patients in this functional class. For most patients this means a combined therapy of available substances according to well defined procedures. Patients whose status remain as "intermediate-risk-status" after receiving a dual therapy over 3-6 months shall undergo a subsequent triple therapy including Selexipag. However, this therapy may not lead to an improvement of the risk-status or even worsened. In these cases, a subcutaneous or intravenous therapy with prostanoids is indicated.

Currently, there are no data available for those patients treated with at least three months with Selexipag as part of a triple therapy that undergo a subsequent intravenous therapy with Treprostinil if there is no change in their risk-status. In the planned study LPS-II, patients are specifically selected on being treated in a dual therapy and having a stagnating intermediate-risk status. These patients receive an implantation of the medical pump LENUS pro, that enables a permanent infusion of Treprostinil.

The aim of this study is to examine, whether patients can reach an improvement in their intermediate-risk-status after six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pulmonary arterial hypertension (WHO group I) accordingly to international guidelines
* intermediate or high risk-profile of PAH after at least three months treatment with vasoactive substances including Selexipag
* indication of intravenous therapy with Treprostinil
* informed consent given for implantation of the medical pump LENUS pro
* informed consent given for participation in the LPS-II study

Exclusion Criteria:

* contraindications according to package information leaflet (LENUS pro) and/or summary of product characteristics (Treprostinil)
* Patient is diagnosed with PAH with an etiology different from that of the inclusion criteria
* chronic kidney insufficiency (estimated GFR < 30)
* hepatic insufficiency: CHILD C (known information from patients medical records)
* intake of substances with potential for infections: intravenous drug abuse, prednisolone, azathioprine, cyclophosphamide
* suffering from diseases with potential for infections: immunodeficiency syndrome, diabetes mellitus, diabetic gangrene
* pregnant or breastfeeding women
* women of childbearing potential who are not on a reliable and safe form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAH (Pulmonary arterial hypertension) who need to undergo treatment with Treprostinil, administered by an intravenous pump system (LENUS pro)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Recovery of clinical stability criteria | Baseline and after 6 months intravenous therapy with Treprostinil
  to achieve "low-risk-status"

SECONDARY OUTCOMES:
Quality of Life | Baseline and after 6 months intravenous therapy with Treprostinil
  Assessment of Quality of Life by EQ-5D-5F questionnaire (patient reported)
Restrictions caused by the implant | immediately after implantation until 6 months intravenous therapy with Treprostinil
  Assessment of restrictions that may cause by the implant: mobility, pain, rubor, swelling
Polysomnography | Baseline and after 6 months intravenous therapy with Treprostinil
  Record of hypnogram: duration of sleep, respiratory analysis, quantity and severity of apnea and hypopnea, snoring, oxygen saturation, heart rate, Continuous Positive Airway Pressure

OTHER OUTCOMES:
Adverse Events associated with the implant | at any visit
  Record of all security related adverse events related to implantation of the pump: infections (local, systemic), seroma/hematoma, dysfunction of the pump, other complications associated with the catheter

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - DRK Kliniken Berlin Westend, Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Gießen, Giessen
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No